CLINICAL TRIAL: NCT03754244
Title: A Phase I Study of TQ-B3456 on Tolerance and Pharmacokinetics
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The enrolment task cannot be gotten within the planned time.It mainly includes patients with non-small cell lung cancer failed in standard treatment,with a short survival period.It is hard to obtain observational endpoints for bone-related events.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3456-I-01
Record Dates: First submitted 2018-11-23; First posted 2018-11-27 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3456 (Experimental): p.o. qd
  Interventions: Drug: TQB3456

INTERVENTIONS:
Drug: TQB3456 — Observe the safety and pk when the subjects take TQB3456 p.o. qd

SUMMARY:
To study the pharmacokinetic characteristics of TQ-B3456 in the human body, recommend a reasonable regimen for subsequent research.

ELIGIBILITY:
Inclusion Criteria:

- progressive or metastatic non-small cell lung cancer that diagnosed Pathologically or cytologically diagnosed patients who have received EGFR tyrosine kinase inhibitor monotherapy (e.g., gefetinib, erlotinib, ecotinib, afatinib) for disease progression EGFR T790M mutation was confirmed ECOG PS≤1 Adequate blood cell counts, kidney function and liver function Patients should participate in the study voluntarily and sign informed consent

Exclusion Criteria:

Patients with non-small-cell lung cancer who have received osimertinib or other raw materials or preparations for EGFRT790M mutant drugs Hypertension (systolic BP ≥140 mmHg, diastolic BP ≥90 mmHg) still uncontrollable by one medication; Hepatitis B virus patients with active replication (DNA> 500 cps / mL), hepatitis C; Patients with immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or organ transplant history

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicities（DLT） | Baseline up to 28 days
  an adverse event cccurring after initiation of TQ-B3456 that met any following criteria：
  1. >=Grade 3 of non-hematology toxicity
  2. Grade 4 hematology toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- No. 241 Huaihai West Road, Xuhui District, Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No